CLINICAL TRIAL: NCT03021681
Title: Huai'an First People 's Hospital,Nanjing Medical University
Brief Title: An Exploratory Study on the Treatment of Chronic Obstructive Pulmonary Disease With Autologous Bronchial Basal Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huai'an No.1 People's Hospital (Other)
Collaborators: Regend Therapeutics (Industry)
Responsible Party: Principal Investigator, ZiLi Meng, Director of respiratory Medicine in Huai'an No.1 People's Hospital, Huai'an No.1 People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Huaian1PH2
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2020-08

CONDITIONS: Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD group(self control) (Other): Prior treatment:20 stable COPD patients were enrolled,estimated the respiratory function and serum index Intervention:autologous bronchial basal cell transplantation After treatment:Estimate the change of respiratory function and serum index in third days , first months, third months, sixth months and first years of the follow-up after treatment respectively
  Interventions: Other: autologous bronchial basal cell transplantation

INTERVENTIONS:
Other: autologous bronchial basal cell transplantation — the investigators obtained extraction bronchial basal cells micro tissue from 3~4 grade bronchus, then purified and selectively amplified bronchial basal cells to reserve . After a period of time, the basal lamina of the bronchial epithelial cells can be stored in the liquid nitrogen cell bank for a long time. Before applied to the patient, bronchial basal cells need to go through a series of strict examination. Then, bronchoscopy was performed again and the bronchial basal lamina suspension was injected directly into the lesion site .

SUMMARY:
Chronic obstructive pulmonary disease(COPD)is characterized by recurrent cough, expectoration and asthma, and eventually develop chronic pulmonary heart disease ,chronic respiratory failure and even death. The current clinical treatments for these patients are symptomatic treatment cannot solve the problem of the damaged lung structure fundamentally. Recent studies show that bronchial basement the layer of cells is a kind of cells in the bronchial epithelial basal layer position, the specific expression of Krt5 antigen with the regeneration and repair of lung function , these cells have the activity similar to adult tissue stem cells. Its division and migration are more active and can continue to produce new cells to complement the death of other types of epithelial cells with functional plasticity which can be used to direct repair the bronchial and alveolar structures. It has been proved that bronchial basal cell transplantation can repair the damaged lungs of experimental animals . The bronchial basal cells from autologous tissue, so there is no immune rejection problem. Also because the bronchial basal cells derived from adult tissues which is a part of the body, so there is no risk of a tumor (in animal experiments, In animal experiments, bronchial basal cells transtracheal input 100 times in human dose still no tumor formation). In the early stage, patients with COPD (2 cases), bronchiectasis (2 cases) and interstitial lung disease (1 case) received the treatment, and the overall effect was good. Diseases were alleviated and recovered to some different extend.The study was to brush bronchial basal cells through fiberbronchoscopy in COPD patients and cultured in vitro, and then through the bronchoscope transfusion to the lesion site. To preliminary evaluate the efficacy and safety of autologous bronchial basal cells in the treatment of chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Between November 2016 and November 2019, the investigators initially recruited 20 with stable COPD patients. Primary evaluations including medical history, physical examination, anthropometric data, blood routine, blood biochemistry, blood coagulation, electrocardiogram,high resolution chest CT, arterial blood gas, pulmonary function test,6-min walking test(6MWT),modified medical research council(MMRC),St George's respiratory questionnaire(SGRQ). After initial evaluation, the investigators obtained extraction bronchial basal cells micro tissue from 3~4 grade bronchus to by mean of fiberbronchoscopy, then purified and selectively amplified bronchial basal cells to reserve .The basal layer cell culture system for our partners (Regend Therapeutics) patented technology using culture medium containing special combination of growth factors and composite materials to simulated composite basal layer environment and can selectively amplified bronchial basal cells, while other types of mature epithelial cells and fibroblasts could not grow naturally. After a period of time, the basal lamina of the bronchial epithelial cells can be stored in the liquid nitrogen cell bank for a long time. Before applied to the patient, bronchial basal cells need to go through a series of strict examination. Then, bronchoscopy was performed again and the bronchial basal lamina suspension was injected directly into the lesion site . Estimate the change of respiratory function(symptoms, signs, chest CT, pulmonary function, the 6 minute walk test, MMRC, SGRQ etc) and serum index in third days , first months, third months, sixth months and first years of the follow-up after treatment respectively, to evaluate the safety and efficiency of autologous bronchial basal cells for treatment of COPD .

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 to 70 years
2. according to the guideline criteria, the diagnosis of COPD:

   ①There is a chronic cough, sputum or gas breathing symptoms such as promoting

   ②Pulmonary function tests showed airflow limitation(FEV1<80% predicted value，FEV1/FVC<0.7)
3. CT imaging and hematological examination excluded other lung diseases.
4. stable disease for more than 2 weeks
5. patients who were able to tolerate fiberoptic bronchoscopy
6. to sign the informed consent form

Exclusion Criteria:

1. women who are pregnant, nursing or not taking effective contraception
2. syphilis, HIV antibody positive person
3. there is a history of alcohol or illicit drug abuse
4. patients who had received any other clinical trial within the first 3 months
5. poor compliance, it is difficult to complete the study
6. researchers believe there may be any increase in the risk of the subject or any interference with the clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11; Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
forced expiratory volume in one second(FEV1) | 24 months
  as the severity of chronic obstructive pulmonary disease(COPD)estimated by pulmonary function
chest high-resolution computed tomography | 24 months
  as the severity of lung hyperinflation estimated by radiological
arterial blood gas | 24 months
  to assess the level of hypoxemia and hypercapnia in chronic obstructive pulmonary disease(COPD) patients
6MWT | 24 months
  6 min walking test, to evaluate the exercise function in patients with moderate and severe pulmonary heart diseases

SECONDARY OUTCOMES:
forced vital capacity(FVC) | 24 months
  an index of pulmonary function in chronic obstructive pulmonary disease(COPD) patients
MMRC | 24 months
  an index to evaluate the lever of dyspnea
SGRQ | 24 months
  a questionnaire to assess the influence of chronic airflow restriction on the quality of life, including symptoms, activities and daily life affected by diseases

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zuo, PhD, Study Chair — Regend Therapeutics,Suzhou Industry Park,Suzhou,CHINA
Locations (1):
- Huai'an First People's Hospital, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuo W, Zhang T, Wu DZ, Guan SP, Liew AA, Yamamoto Y, Wang X, Lim SJ, Vincent M, Lessard M, Crum CP, Xian W, McKeon F. p63(+)Krt5(+) distal airway stem cells are essential for lung regeneration. Nature. 2015 Jan 29;517(7536):616-20. doi: 10.1038/nature13903. Epub 2014 Nov 12. PMID 25383540
- [Background] Kumar PA, Hu Y, Yamamoto Y, Hoe NB, Wei TS, Mu D, Sun Y, Joo LS, Dagher R, Zielonka EM, Wang de Y, Lim B, Chow VT, Crum CP, Xian W, McKeon F. Distal airway stem cells yield alveoli in vitro and during lung regeneration following H1N1 influenza infection. Cell. 2011 Oct 28;147(3):525-38. doi: 10.1016/j.cell.2011.10.001. PMID 22036562
- [Background] Rock JR, Randell SH, Hogan BL. Airway basal stem cells: a perspective on their roles in epithelial homeostasis and remodeling. Dis Model Mech. 2010 Sep-Oct;3(9-10):545-56. doi: 10.1242/dmm.006031. Epub 2010 Aug 10. PMID 20699479